A single center randomized prospective study on the peristaltic direction of gastrointestinal anastomosis in Roux-en-Y reconstruction after distal curative gastrectomy for gastric cancer (DJY002 Trail)

**Edition Number: 1.0** 

**Edition Generation Date: Qct 30, 2020** 

Principal Investigator: Jingyu Deng and Han Liang

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## **Protocol:**

- Distal gastric adenocarcinoma (antrum, pylorus, angle, and/or lower part of body) identified by histopathologic examination without non-curative resection factors
- Undergo potentially curative gastrectomy plus lymphadenectomy (cTanyNanyM0)
- Age between 18 and 70 years
- KPS score >60
- No neoadjuvant therapy
- No seriously chronic diseases of important organs



after distal curative gastrectomy for gastric cancer.